CLINICAL TRIAL: NCT01824849
Title: The Comparison of Voice and Swallowing Parameters After Endoscopic Total and Partial Arytenoidectomy Using Medially Based Mucosal Advancement Flap Technique for Bilateral Abductor Vocal Fold Paralysis: A Randomized Trial
Brief Title: Total Versus Partial Arytenoidectomy in Bilateral Vocal Fold Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Taner Yilmaz, Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUmedTY1
Record Dates: First submitted 2013-03-28; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Airway Obstruction; Vocal Cord Paralysis
Keywords: Vocal cords; Vocal cord paralysis; Arytenoid cartilage
MeSH Terms: conditions — Airway Obstruction; Vocal Cord Paralysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total arytenoidectomy (Experimental): Endoscopic total arytenoidectomy was performed on patients.
  Interventions: Procedure: Total arytenoidectomy
- Partial arytenoidectomy (Experimental): Endoscopic partial arytenoidectomy was performed on patients.
  Interventions: Procedure: Partial arytenoidectomy

INTERVENTIONS:
Procedure: Total arytenoidectomy — Endoscopic total arytenoidectomy was performed on patients with bilateral vocal fold paralysis
  Arms: Total arytenoidectomy
Procedure: Partial arytenoidectomy — Endoscopic partial arytenoidectomy was performed on patients with bilateral vocal fold paralysis
  Arms: Partial arytenoidectomy

SUMMARY:
Total arytenoidectomy is claimed to increase risk of aspiration and cause more voice loss than other operations performed for bilateral vocal fold paralysis (BVFP). However, objective evidence for such conclusion is lacking. There is no study comparing swallowing and voice after total and partial arytenoidectomy.

DETAILED DESCRIPTION:
Design: Prospective, randomized, double-blind, case-control Setting: Tertiary, referral, university Patients: Twenty patients with BVFP Intervention: Endoscopic total and partial arytenoidectomy

ELIGIBILITY:
Inclusion Criteria:

* Bilateral vocal fold paralysis

Exclusion Criteria:

* Previously operated patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Decannulation | From the day of operation until 52 weeks after arytenoidectomy
  Preoperative examinations were repeated 1 year after surgery.

SECONDARY OUTCOMES:
Duration of operation | At the day of operation
  The duration of operation was measured in minutes at the day of operation.

OTHER OUTCOMES:
Voice Handicap Index | From the day of operation until 52 weeks after arytenoidectomy
  Voice Handicap Index is a 30-item questionnaire. Possible points change between 0 to 120. Zero means normal voice, 120 means the worst voice. Preoperative examinations were repeated 1 year after surgery.
Acoustic analysis | From the day operation until 52 weeks after arytenoidectomy
  Fundamental frequency (Hertz), absolute jitter (microseconds), shimmer percent (%), noise to harmonic ratio will be measured as physical measures of voice.
Aerodynamic analysis | From the day of operation until 52 weeks after arytenoidectomy
  Maximum phonation time (seconds), mean flow rate (liters/second), mean resistance (cmH20/liter/second), mean power (Watt), mean efficiency (ppm) and mean pressure (cmH2O)are obtained as physical measures of aerodynamic analysis.
Postoperative breathing ability | 52 weeks after arytenoidectomy
  Breathing ability was evaluated on a scale of -2 to +2 (-2: significantly worse; -1: somewhat worse; 0: no change; +1: somewhat better; +2: significantly better).
Subjective comparison of pre- and postoperative voice by a phoniatrician | From the day of operation until 52 weeks after arytenoidectomy
  Subjective comparison of pre- and postoperative voice on a scale of -2 to +2 (-2: significantly worse; -1: somewhat worse; 0: no change; +1: somewhat better; +2: significantly better).
Speech intensity | 52 weeks after arytenoidectomy
  Speech intensity is measured in decibels.
Functional outcome swallowing scale | 52 weeks after arytenoidectomy
  Functional Outcome Swallowing Scale: 0-5 (0: Normal function and asymptomatic; 1: Normal function with episodic or daily symptoms of dysphagia; 2: Compensated abnormal function manifested by significant dietary modifications or prolonged mealtime (without weight loss or aspiration); 3: Decompensated abnormal function with weight loss of <10% of body weight over 6 months due to dysphagia; or daily cough, gagging or aspiration during meals; 4: Severely decompensated abnormal function with weight loss of >10% of body weight over 6 months due to dysphagia; or severe aspiration with bronchopulmonary complications. Non oral feeding for most nutrition; 5: Non oral feeding for all nutrition).

CONTACTS AND LOCATIONS:
Overall Officials: Taner Yilmaz, MD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Yilmaz T. Endoscopic total arytenoidectomy for bilateral abductor vocal fold paralysis: a new flap technique and personal experience with 50 cases. Laryngoscope. 2012 Oct;122(10):2219-26. doi: 10.1002/lary.23467. Epub 2012 Aug 2. PMID 22865083
- [Background] Dursun G, Gokcan MK. Aerodynamic, acoustic and functional results of posterior transverse laser cordotomy for bilateral abductor vocal fold paralysis. J Laryngol Otol. 2006 Apr;120(4):282-8. doi: 10.1017/S0022215106000715. PMID 16623972
- [Background] THORNELL WC. Transoral intralaryngeal approach for arytenoidectomy in bilateral vocal cord paralysis with inadequate airway. Ann Otol Rhinol Laryngol. 1957 Jun;66(2):364-8. No abstract available. PMID 13459231
- [Background] Sapundzhiev N, Lichtenberger G, Eckel HE, Friedrich G, Zenev I, Toohill RJ, Werner JA. Surgery of adult bilateral vocal fold paralysis in adduction: history and trends. Eur Arch Otorhinolaryngol. 2008 Dec;265(12):1501-14. doi: 10.1007/s00405-008-0665-1. Epub 2008 Apr 17. PMID 18418622
- [Background] Kleinsasser O, Nolte E. [Report on the indication, technique and functional results of endolaryngeal arytenoidectomy and submucous partial chordectomy in bilateral paralysis of vocal cord (author's transl)]. Laryngol Rhinol Otol (Stuttg). 1981 Aug;60(8):397-401. German. PMID 7346673
- [Background] Remacle M, Lawson G, Mayne A, Jamart J. Subtotal carbon dioxide laser arytenoidectomy by endoscopic approach for treatment of bilateral cord immobility in adduction. Ann Otol Rhinol Laryngol. 1996 Jun;105(6):438-45. doi: 10.1177/000348949610500604. PMID 8638894
- [Background] Salassa JR. A functional outcome swallowing scale for staging oropharyngeal dysphagia. Dig Dis. 1999;17(4):230-4. doi: 10.1159/000016941. PMID 10754363
- [Background] Plouin-Gaudon I, Lawson G, Jamart J, Remacle M. Subtotal carbon dioxide laser arytenoidectomy for the treatment of bilateral vocal fold immobility: long-term results. Ann Otol Rhinol Laryngol. 2005 Feb;114(2):115-21. doi: 10.1177/000348940511400206. PMID 15757190
- [Background] Crumley RL. Endoscopic laser medial arytenoidectomy for airway management in bilateral laryngeal paralysis. Ann Otol Rhinol Laryngol. 1993 Feb;102(2):81-4. doi: 10.1177/000348949310200201. PMID 8427504
- [Background] Bosley B, Rosen CA, Simpson CB, McMullin BT, Gartner-Schmidt JL. Medial arytenoidectomy versus transverse cordotomy as a treatment for bilateral vocal fold paralysis. Ann Otol Rhinol Laryngol. 2005 Dec;114(12):922-6. doi: 10.1177/000348940511401205. PMID 16425557
- [Background] Young VN, Rosen CA. Arytenoid and posterior vocal fold surgery for bilateral vocal fold immobility. Curr Opin Otolaryngol Head Neck Surg. 2011 Dec;19(6):422-7. doi: 10.1097/MOO.0b013e32834c1f1c. PMID 21986801
- [Background] Hillel AD, Benninger M, Blitzer A, Crumley R, Flint P, Kashima HK, Sanders I, Schaefer S. Evaluation and management of bilateral vocal cord immobility. Otolaryngol Head Neck Surg. 1999 Dec;121(6):760-5. doi: 10.1053/hn.1999.v121.a98733. PMID 10580234
- [Derived] Yilmaz T, Suslu N, Atay G, Ozer S, Gunaydin RO, Bajin MD. Comparison of voice and swallowing parameters after endoscopic total and partial arytenoidectomy for bilateral abductor vocal fold paralysis: a randomized trial. JAMA Otolaryngol Head Neck Surg. 2013 Jul;139(7):712-8. doi: 10.1001/jamaoto.2013.3395. PMID 23868428